CLINICAL TRIAL: NCT05173012
Title: A Phase 2, Double-Blind, Randomized, Placebo-Controlled, Dose-Response Study of SAGE-324 for the Treatment of Essential Tremor
Brief Title: Study to Evaluate SAGE-324 in Participants With Essential Tremor
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sage Therapeutics (Industry)
Collaborators: Biogen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 324-ETD-202
Record Dates: First submitted 2021-12-15; First posted 2021-12-29 (Actual); Results first posted 2025-05-16 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-05

CONDITIONS: Essential Tremor
Keywords: Essential Tremor; SAGE-324
MeSH Terms: conditions — Essential Tremor

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- SAGE-324 Matched Placebo (Placebo Comparator): Participants will receive SAGE-324 matched placebo, stratified by baseline propranolol use.
  Monotherapy:
  Participants will receive SAGE-324 matched placebo, oral tablets, once daily (QD), in the evening, from Day 1 to Day 90 in a double-blind treatment period.
  Adjunct therapy:
  Participants will receive SAGE-324 matched placebo, oral tablets, QD, in the evening, from Day 1 to Day 90 along with a stable dose of up to 320 milligrams (mg) of propranolol from 3 months prior to Screening up to Day 90 in a double-blind treatment period.
  Interventions: Drug: SAGE-324 Matched Placebo
- SAGE-324 15 mg (Experimental): Participants will receive SAGE-324, 15 mg, stratified by baseline propranolol use.
  Monotherapy:
  Participants will receive SAGE-324, 15 mg, oral tablets, QD, in the evening, from Day 1 to Day 90 in a double-blind treatment period.
  Adjunct therapy:
  Participants will receive SAGE-324, 15 mg, oral tablets, QD, in the evening, from Day 1 to Day 90 along with a stable dose of up to 320 mg of propranolol from 3 months prior to Screening up to Day 90 in a double-blind treatment period.
  Interventions: Drug: SAGE-324
- SAGE-324 30 mg (Experimental): Participants will receive SAGE-324, 30 mg, stratified by baseline propranolol use.
  Monotherapy:
  Participants will receive SAGE-324, 30 mg, oral tablets, QD, in the evening, from Day 1 to Day 90 in a double-blind treatment period.
  Adjunct therapy:
  Participants will receive SAGE-324, 30 mg, oral tablets, QD, in the evening, from Day 1 to Day 90 along with a stable dose of up to 320 mg of propranolol from 3 months prior to Screening up to Day 90 in a double-blind treatment period.
  Interventions: Drug: SAGE-324
- SAGE-324 60 mg (Experimental): Participants will receive SAGE-324: 15 mg, 30 mg, 45 mg, and 60 mg, stratified by baseline propranolol use.
  Monotherapy:
  Participants will receive SAGE-324, 15 mg from Day 1 to 14, followed by up-titration to 30 mg from Day 15 to 28, then to 45 mg from Day 29 to 42, and then to 60 mg from Day 43 to 90, oral tablets, QD, in the evening, from Day 1 to Day 90 in a double-blind treatment period.
  Adjunct therapy:
  Participants will receive SAGE-324, 15 mg from Day 1 to 14, followed by up-titration to 30 mg from Day 15 to 28, then to 45 mg from Day 29 to 42, and then to 60 mg from Day 43 to 90, oral tablets, QD, in the evening, from Day 1 to Day 90 along with a stable dose of up to 320 mg of propranolol from 3 months prior to Screening up to Day 90 in a double-blind treatment period.
  Interventions: Drug: SAGE-324

INTERVENTIONS:
Drug: SAGE-324 — SAGE-324 oral tablets.
  Arms: SAGE-324 15 mg; SAGE-324 30 mg; SAGE-324 60 mg
Drug: SAGE-324 Matched Placebo — SAGE-324 matched placebo oral tablets.
  Arms: SAGE-324 Matched Placebo

SUMMARY:
The primary purpose of this study is to evaluate the dose-response relationship of different doses of SAGE-324 on upper extremity tremor in participants with essential tremor (ET) in the monotherapy cohort.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of ET, as defined by all of the following criteria:

   * Isolated tremor syndrome consisting of bilateral upper limb action tremor
   * At least 3 years duration
   * With or without tremor in other locations (eg, head, voice, or lower limbs)
2. Absence of other neurological signs, such as dystonia, ataxia, or parkinsonism, isolated focal tremors (eg, voice, head), task- and position-specific tremors, sudden tremor onset, or evidence of stepwise deterioration of tremor.
3. Participant has the following:

   * Scores of at least 12 in the combined TETRAS Performance Subscale Item 4 (upper limb tremor) at both Screening and pre-dose on Day 1
   * Scores of at least 6 in the total TETRAS Performance Subscale Item 4 score for the dominant upper limb (the sum of the three items for either the right or left upper limb, whichever is dominant) at both Screening and pre-dose on Day 1
4. Participant has a baseline TETRAS ADL Subscale score of at least 20 at Screening.
5. Willing to discontinue medications taken for the treatment of ET except propranolol at least 14 days or 5 half-lives (whichever is longer) prior to receiving the investigational product (IP). Medications taken for the treatment of ET that were discontinued prior to receiving IP may be resumed following Day 97. Participants in the adjunct therapy cohort must be on a stable dose of propranolol (maximum total daily propranolol dose up to 320 mg allowed) for the treatment of ET from 3 months prior to Screening through Day 97 of the study.
6. Participant is willing to limit use of alcohol to 2 units per day for males and 1 unit per day for females starting at least 1 week prior to Day 1 and through Day 97 of the study.
7. Participant is willing to maintain prestudy consumption of products that contain nicotine starting at least 1 week prior to Day 1 and through Day 97 of the study.

Exclusion Criteria:

1. Presence of known causes of enhanced physiological tremor.
2. Participant has had newly administered tremorgenic drugs (14 days or 5 half-lives [whichever is longer] prior to Day 1) or presence of alcohol withdrawal state.
3. Direct or indirect injury or trauma to the nervous system within 3 months before the onset of tremor.
4. Previous procedure for the treatment of ET, deep brain stimulation, brain lesioning, or magnetic resonance (MR) guided procedure, eg, MR-guided focused ultrasound. Use of Cala Trio bracelet for the treatment of ET from two weeks prior to Day 1 through Day 97 is prohibited.
5. Participant has had botulinum toxin for treatment of ET within 6 months of Screening.
6. Historical or clinical evidence of tremor with functional neurological syndrome origin.
7. Participant currently requires propranolol treatment for a medical condition other than ET.
8. Participant has history of substance abuse or dependence prior to Screening, has a positive screen for drugs of abuse at Screening or predose on Day 1. Participants with nicotine use disorder that impacts their tremor are excluded.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 146 (Actual)
Dates: Start 2022-01-05 (Actual); Primary Completion 2024-05-02 (Actual); Study Completion 2024-05-16 (Actual)

CONTACTS AND LOCATIONS:
Locations (48):
- United States (48):
  - Sage Investigational Site, Hoover, Alabama
  - Sage Investigational Site, Phoenix, Arizona
  - Sage Investigational Site, Scottsdale, Arizona
  - Sage Investigational Site, Sun City, Arizona
  - Sage Investigational Site, Fountain Valley, California
  - Sage Investigational Site, Fullerton, California
  - Sage Investigational Site, Los Angeles, California
  - Sage Investigational Site, Englewood, Colorado
  - Sage Investigational Site, Boca Raton, Florida
  - Sage Investigational Site, Boynton Beach, Florida
  - Sage Investigational Site, Bradenton, Florida
  - Sage Investigational Site, Coral Springs, Florida
  - Sage Investigational Site, Gainesville, Florida
  - Sage Investigational Site, Hollywood, Florida
  - Sage Investigational Site, Kendall, Florida
  - Sage Investigational Site, Miami, Florida
  - Sage Investigational Site, Naples, Florida
  - Sage Investigational Site, Orlando, Florida
  - Sage Investigational Site, Pensacola, Florida
  - Sage Investigational Site, Port Charlotte, Florida
  - Sage Investigational Site, Tampa, Florida
  - Sage Investigational Site, Atlanta, Georgia
  - Sage Investigational Site, Decatur, Georgia
  - Sage Investigational Site, Chicago, Illinois
  - Sage Investigational Site, Springfield, Illinois
  - Sage Investigational Site, Kansas City, Kansas
  - Sage Investigational Site, Lexington, Kentucky
  - Sage Investigational Site, Shreveport, Louisiana
  - Sage Investigational Site, Boston, Massachusetts
  - Sage Investigational Site, Farmington Hills, Michigan
  - Sage Investigational Site, Lansing, Michigan
  - Sage Investigational Site, Las Vegas, Nevada
  - Sage Investigational Site, New York, New York
  - Sage Investigational Site, Asheville, North Carolina
  - Sage Investigational Site, Cincinnati, Ohio
  - Sage Investigational Site, Dayton, Ohio
  - Sage Investigational Site, Tulsa, Oklahoma
  - Sage Investigational Site, Memphis, Tennessee
  - Sage Investigational Site, Austin, Texas
  - Sage Investigational Site, Fort Worth, Texas
  - Sage Investigational Site, Houston, Texas
  - Sage Investigational Site, Katy, Texas
  - Sage Investigational Site, Round Rock, Texas
  - Sage Investigational Site, San Antonio, Texas
  - Sage Investigational Site, McLean, Virginia
  - Sage Investigational Site, West Falls Church, Virginia
  - Sage Investigational Site, Kirkland, Washington
  - Sage Investigational Site, Spokane, Washington

IPD SHARING:
Plan to Share IPD: No
Data sharing will be consistent with the results submission policy of ClinicalTrials.gov.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at 51 investigative sites in the United States from 05 Jan 2022 to 16 May 2024.
Pre-assignment Details: A total of 160 participants were planned for the study, of which 147 participants were randomized. Out of 147, 1 participant was randomized in error but was not assigned in any of the treatment group. This participant did not receive any treatment, therefore only146 participants received IP.
Groups:
- Monotherapy: Placebo: Participants received SAGE-324 matched placebo, orally, once daily (QD), in the evening, from Day 1 to Day 90 in a double-blind treatment period.
- Monotherapy: SAGE-324 15 mg: Participants received SAGE-324 15 milligrams (mg), orally, QD, in the evening, from Day 1 to Day 90 in a double-blind treatment period.
- Monotherapy: SAGE-324 30 mg: Participants received SAGE-324 30 mg, orally, QD, in the evening, from Day 1 to Day 90 in a double-blind treatment period.
- Monotherapy: SAGE-324 60 mg: Participants received SAGE-324 15 mg from Day 1 to 14, followed by up-titration to 30 mg from Day 15 to 28, then to 45 mg from Day 29 to 42, and then to 60 mg from Day 43 to 90, orally, QD, in the evening, from Day 1 to Day 90 in a double-blind treatment period.
- Adjunct Therapy: Placebo: Participants received SAGE-324 matched placebo, orally, QD, in the evening, from Day 1 to Day 90 along with a stable dose of up to 320 mg of propranolol from 3 months prior to screening up to Day 90 in a double-blind treatment period.
- Adjunct Therapy: SAGE-324 15 mg: Participants received SAGE-324 15 mg, orally, QD, in the evening, from Day 1 to Day 90 along with a stable dose of up to 320 mg of propranolol from 3 months prior to Screening up to Day 90 in a double-blind treatment period.
- Adjunct Therapy: SAGE-324 30 mg: Participants received SAGE-324, 30 mg orally, QD, in the evening, from Day 1 to Day 90 along with a stable dose of up to 320 mg of propranolol from 3 months prior to Screening up to Day 90 in a double-blind treatment period.
- Adjunct Therapy: SAGE-324 60 mg: Participants received SAGE-324, 15 mg from Day 1 to 14, followed by up-titration to 30 mg from Day 15 to 28, then to 45 mg from Day 29 to 42, and then to 60 mg from Day 43 to 90, orally, QD, in the evening along with a stable dose of up to 320 mg of propranolol from 3 months prior to Screening up to Day 90 in a double-blind treatment period.
Period: Overall Study
Arm/Group | Monotherapy: Placebo | Monotherapy: SAGE-324 15 mg | Monotherapy: SAGE-324 30 mg | Monotherapy: SAGE-324 60 mg | Adjunct Therapy: Placebo | Adjunct Therapy: SAGE-324 15 mg | Adjunct Therapy: SAGE-324 30 mg | Adjunct Therapy: SAGE-324 60 mg
Started | 31 | 32 | 32 | 33 | 4 | 4 | 5 | 5
Completed | 28 | 29 | 27 | 13 | 3 | 4 | 2 | 1
Not Completed | 3 | 3 | 5 | 20 | 1 | 0 | 3 | 4
Not completed — Adverse Event | 2 | 3 | 4 | 13 | 0 | 0 | 2 | 4
Not completed — Lost to Follow-up | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 1 | 3 | 1 | 0 | 1 | 0
Not completed — Protocol Deviation | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Other | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The Safety Analysis Set included all participants who were administered investigational product (IP).
Groups:
- Monotherapy: Placebo: Participants received SAGE-324 matched placebo, orally, QD, in the evening, from Day 1 to Day 90 in a double-blind treatment period.
- Monotherapy: SAGE-324 15 mg: Participants received SAGE-324 15 mg, orally, QD, in the evening, from Day 1 to Day 90 in a double-blind treatment period.
- Adjunct Therapy: SAGE-324 15 mg: Participants received SAGE-324 15 mg, oral tablets, QD, in the evening, from Day 1 to Day 90 along with a stable dose of up to 320 mg of propranolol from 3 months prior to screening up to Day 90 in a double-blind treatment period.
- Adjunct Therapy: SAGE-324 60 mg: Participants received SAGE-324, 15 mg from Day 1 to 14, followed by up-titration to 30 mg from Day 15 to 28, then to 45 mg from Day 29 to 42, and then to 60 mg from Day 43 to 90, oral tablets, QD, in the evening, from Day 1 to Day 90 along with a stable dose of up to 320 mg of propranolol from 3 months prior to screening up to Day 90 in a double-blind treatment period.
- Total: Total of all reporting groups
Arm/Group | Monotherapy: Placebo | Monotherapy: SAGE-324 15 mg | Monotherapy: SAGE-324 30 mg | Monotherapy: SAGE-324 60 mg | Adjunct Therapy: Placebo | Adjunct Therapy: SAGE-324 15 mg | Adjunct Therapy: SAGE-324 30 mg | Adjunct Therapy: SAGE-324 60 mg | Total
Number analyzed (Participants) | 31 | 32 | 32 | 33 | 4 | 4 | 5 | 5 | 146
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.3 (9.35) | 65.8 (11.25) | 66.9 (10.18) | 69.5 (7.67) | 65.8 (11.95) | 69.3 (11.59) | 67.4 (7.57) | 69.8 (8.87) | 67.9 (9.60)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 11 | 10 | 14 | 1 | 2 | 2 | 3 | 54
  Male | 20 | 21 | 22 | 19 | 3 | 2 | 3 | 2 | 92
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 1 | 4 | 0 | 0 | 0 | 0 | 7
  Not Hispanic or Latino | 30 | 31 | 31 | 29 | 4 | 4 | 5 | 5 | 139
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 2 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 4
  White | 29 | 32 | 30 | 31 | 3 | 4 | 5 | 5 | 139
  More than one race | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
The Essential Tremor Rating Assessment Scale (TETRAS) Performance Subscale Item 4 (Upper Limb) Score [Mean (Standard Deviation); unit: score on a scale] — TETRAS is clinical evaluation of essential tremor. For the TETRAS Performance Subscale Item 4 (upper limb), three maneuvers/assessments were to be completed for both arms, first for right arm and then for left, specifically Item 4a, limbs extended forward maneuver (postural tremor), Item 4b, wing-beating [elbows flexed] maneuver (postural tremor), & Item 4c finger-nose-finger maneuver (kinetic tremor). Each item score ranges from 0 to 4; with 0 to 12 being the score range for each arm of body. Total upper limb score combined for both arms range from 0 to 24. Higher scores=more severe tremor. Population: The Full Analysis Set included all randomized participants who received any amount of IP and had a baseline and at least one post-baseline TETRAS Performance Subscale Item 4 (upper limb tremor) total score. The number analyzed indicates the number of participants with data available for analysis.
  score on a scale
    number analyzed (Participants) | 31 | 32 | 31 | 33 | 4 | 4 | 5 | 5 | 145
    (all) | 13.68 (1.249) | 13.69 (1.430) | 13.10 (1.625) | 13.39 (1.633) | 12.50 (0.577) | 14.25 (2.843) | 13.20 (0.758) | 13.00 (0.935) | 13.43 (1.492)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in The Essential Tremor Rating Assessment Scale (TETRAS) Performance Subscale Item 4 (Upper Limb) Total Score on Day 91 in the Monotherapy Cohort
Description: TETRAS is a clinical evaluation of essential tremor. The TETRAS performance subscale upper limb tremor score is a component of TETRAS. For the TETRAS Performance Subscale Item 4 (upper limb), three maneuvers/assessments were to be completed for both arms, first for the right arm and then for the left, specifically Item 4a, limbs extended forward maneuver (postural tremor), Item 4b, wing-beating [elbows flexed] maneuver (postural tremor), and Item 4c finger-nose-finger maneuver (kinetic tremor). Each assessment is rated on a 0 to 4 scale of severity in 0.5-point increments, with higher scores indicating more severe tremor. The Performance Subscale Item 4 (upper limb) total score range for a given side (left or right) is 0 to 12, and for both sides combined is 0 to 24. A negative change from baseline indicates improvement. Mixed model for repeated measures (MMRM) was used for the analysis.
Time Frame: Baseline, Day 91
Population: The Full Analysis Set included all randomized participants who received any amount of IP and had a baseline and at least one post-baseline TETRAS Performance Subscale Item 4 (upper limb tremor) total score. The overall number of participants analyzed indicates the number of participants with data available for outcome measure analysis.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Monotherapy: Placebo | Monotherapy: SAGE-324 15 mg | Monotherapy: SAGE-324 30 mg | Monotherapy: SAGE-324 60 mg
Number analyzed (Participants) | 28 | 28 | 27 | 13
score on a scale | -2.53 (0.445) | -2.14 (0.436) | -2.81 (0.449) | -1.51 (0.540)
Statistical Analysis 1: Comparison: Monotherapy: Placebo vs Monotherapy: SAGE-324 15 mg; Test type: Superiority; p = 0.5325, MMRM; MMRM model included treatment, baseline score, assessment timepoint, and timepoint-by-treatment as explanatory variables, treated as fixed effects; Least Squares (LS) Mean Difference = 0.39, 95% CI 2-sided [-0.84 to 1.62], Standard Error of Mean 0.623 — Difference was calculated as Monotherapy: SAGE-324 15 mg - placebo
Statistical Analysis 2: Comparison: Monotherapy: Placebo vs Monotherapy: SAGE-324 30 mg; Test type: Superiority; p = 0.6549, MMRM; [statistical method as in outcome 1, analysis 1]; LS Mean Difference = -0.28, 95% CI 2-sided [-1.54 to 0.97], Standard Error of Mean 0.634 — Difference was calculated as Monotherapy: SAGE-324 30 mg - placebo
Statistical Analysis 3: Comparison: Monotherapy: Placebo vs Monotherapy: SAGE-324 60 mg; Test type: Superiority; p = 0.1462, MMRM; [statistical method as in outcome 1, analysis 1]; LS Mean Difference = 1.02, 95% CI 2-sided [-0.36 to 2.41], Standard Error of Mean 0.700 — Difference was calculated as Monotherapy: SAGE-324 60 mg - placebo

2. Secondary Outcome: Change From Baseline in TETRAS Activities of Daily Living (ADL) Composite Score in the Monotherapy Cohort
Description: TETRAS ADL Subscale (items 1-12) assesses how ET affects typical ADL (speech, eating, drinking, dressing, personal hygiene, writing, occupational impairment, social impact, activities affected by UL tremor). TETRAS ADL composite score comprises Items 1-11 of ADL Subscale (Item 1: speech impairment; Item 10: occupational impairment; remaining 9 items: impairment in activities affected by UL tremor) and Item 6 of Performance Subscale (spiral drawing). Each of individual item is rated on a scale from 0 (normal activity) to 4 (severe abnormality); responses of 0 & 1 in TETRAS ADL Subscale Items 1 to 11 were collapsed such that scale is 0 (normal/slightly abnormal), 1 (mildly abnormal), 2 (moderately abnormal), and 3 (severely abnormal). Performance Subscale Item 6 responses were collapsed with responses having 0.5 point increments grouped with next higher integer response. ADL composite score range is 0 to 39. Higher score=greater abnormality, negative change=improvement.
Time Frame: Baseline, Day 91
Population: The Full Analysis Set included all randomized participants who received any amount of IP and had a baseline and at least one post-baseline TETRAS Performance Subscale Item 4 (upper limb tremor) total score. The overall number of participants analyzed indicates the number of participants with data available for analysis at specified timepoint.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Monotherapy: Placebo | Monotherapy: SAGE-324 15 mg | Monotherapy: SAGE-324 30 mg | Monotherapy: SAGE-324 60 mg
Number analyzed (Participants) | 28 | 28 | 27 | 13
score on a scale | -4.51 (0.951) | -2.48 (0.921) | -5.29 (0.948) | -3.51 (1.080)
Statistical Analysis 1: Comparison: Monotherapy: Placebo vs Monotherapy: SAGE-324 15 mg; Test type: Superiority; p = 0.1271, MMRM; [statistical method as in outcome 1, analysis 1]; LS Mean Difference = 2.04, 95% CI 2-sided [0.59 to 4.67], Standard Error of Mean 1.326
Statistical Analysis 2: Comparison: Monotherapy: Placebo vs Monotherapy: SAGE-324 30 mg; Test type: Superiority; p = 0.5642, MMRM; [statistical method as in outcome 1, analysis 1]; LS Mean Difference = -0.78, 95% CI 2-sided [-3.45 to 1.89], Standard Error of Mean 1.347
Statistical Analysis 3: Comparison: Monotherapy: Placebo vs Monotherapy: SAGE-324 60 mg; Test type: Superiority; p = 0.4860, MMRM; [statistical method as in outcome 1, analysis 1]; LS Mean Difference = 1.01, 95% CI 2-sided [-1.84 to 3.85], Standard Error of Mean 1.439

ADVERSE EVENTS:
Time Frame: Up to Day 104
Description: The Safety Analysis Set included all participants who were administered IP.
Arm/Group | Monotherapy: Placebo | Monotherapy: SAGE-324 15 mg | Monotherapy: SAGE-324 30 mg | Monotherapy: SAGE-324 60 mg | Adjunct Therapy: Placebo | Adjunct Therapy: SAGE-324 15 mg | Adjunct Therapy: SAGE-324 30 mg | Adjunct Therapy: SAGE-324 60 mg
All-Cause Mortality (participants affected / at risk) | 0/31 | 0/32 | 0/32 | 0/33 | 0/4 | 0/4 | 0/5 | 0/5
Serious Adverse Events (participants affected / at risk) | 1/31 | 1/32 | 0/32 | 1/33 | 0/4 | 0/4 | 1/5 | 0/5
Other Adverse Events (participants affected / at risk) | 9/31 | 13/32 | 15/32 | 22/33 | 1/4 | 3/4 | 3/5 | 5/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Monotherapy: Placebo (N=31) | Monotherapy: SAGE-324 15 mg (N=32) | Monotherapy: SAGE-324 30 mg (N=32) | Monotherapy: SAGE-324 60 mg (N=33) | Adjunct Therapy: Placebo (N=4) | Adjunct Therapy: SAGE-324 15 mg (N=4) | Adjunct Therapy: SAGE-324 30 mg (N=5) | Adjunct Therapy: SAGE-324 60 mg (N=5)
Staphylococcal infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Transient ischaemic attack (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Monotherapy: Placebo (N=31) | Monotherapy: SAGE-324 15 mg (N=32) | Monotherapy: SAGE-324 30 mg (N=32) | Monotherapy: SAGE-324 60 mg (N=33) | Adjunct Therapy: Placebo (N=4) | Adjunct Therapy: SAGE-324 15 mg (N=4) | Adjunct Therapy: SAGE-324 30 mg (N=5) | Adjunct Therapy: SAGE-324 60 mg (N=5)
Somnolence (Nervous system disorders) | 1 | 5 | 8 | 8 | 0 | 0 | 0 | 1
Dizziness (Nervous system disorders) | 0 | 1 | 5 | 6 | 0 | 0 | 0 | 0
Balance disorder (Nervous system disorders) | 0 | 0 | 1 | 5 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 1 | 3 | 0 | 2 | 0 | 1 | 1 | 0
Memory impairment (Nervous system disorders) | 0 | 1 | 0 | 3 | 0 | 0 | 0 | 0
Paraesthesia (Nervous system disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 0 | 3 | 3 | 4 | 0 | 0 | 1 | 2
Feeling abnormal (General disorders) | 0 | 0 | 2 | 4 | 0 | 0 | 1 | 0
Nasopharyngitis (Infections and infestations) | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 0 | 3 | 1 | 0 | 0 | 0 | 0
Abnormal dreams (Psychiatric disorders) | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 1 | 0 | 1 | 2 | 0 | 0 | 0 | 0
Depression (Psychiatric disorders) | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypotension (Vascular disorders) | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Hypertension (Vascular disorders) | 3 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Erectile dysfunction (Reproductive system and breast disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Aphasia (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Cognitive disorder (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Slow speech (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
COVID-19 (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 1
Gastroenteritis viral (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Mouth ulceration (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Gait disturbance (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Head injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Procedural pain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Blood alkaline phosphatase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Blood urea increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Blood bilirubin unconjugated increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Blood thyroid stimulating hormone increased (Investigations) | 2 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Gamma-glutamyltransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Platelet count decreased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Heart rate increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Conjunctival hyperaemia (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Visual acuity reduced (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Apathy (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Glycosuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dyspnoea (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Orthostatic hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The PI can either be a party and subject to the same restrictions as the institution, or if not a party, the restrictions are described on the face of the contract (i.e., PI is a contractor of the institution; PI is part of a larger group of study personnel; institution has contracted with or otherwise bound all study personnel under confidentiality obligations and requirements to vest intellectual property to the institution).

DOCUMENTS (2):
  • Study Protocol (2023-11-08): https://cdn.clinicaltrials.gov/large-docs/12/NCT05173012/Prot_000.pdf
  • Statistical Analysis Plan (2024-06-18): https://cdn.clinicaltrials.gov/large-docs/12/NCT05173012/SAP_001.pdf